CLINICAL TRIAL: NCT02022033
Title: BrUOG 295:Adjuvant FOLFOX-A For Resected Pancreatic Cancer: A Phase II Brown University Oncology Research Group Trial
Brief Title: BrUOG 295: Adjuvant FOLFOX-A For Resected Pancreatic Cancer: A Phase II Brown University Oncology Research Group Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 295
Record Dates: First submitted 2013-11-27; First posted 2013-12-27 (Estimated); Results first posted 2021-09-08 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Adjuvant; Pancreas; Resected; Invasive adenocarcinoma; adenosquamous cancer; Intraductal papillary mucinous neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOXA (Experimental): Abraxane: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.
  Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)
  Interventions: Drug: FOLFOXA

INTERVENTIONS:
Drug: FOLFOXA — Abraxane: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.
  Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)

SUMMARY:
The investigators preliminary data suggests that FOLFOX-A may have equal or superior activity as compared to FOLFIRINOX and appears to be better tolerated. Therefore, FOLFOX-A may be a better regimen in the adjuvant setting for patients with resected pancreatic cancer. This protocol will obtain preliminary data on safety and disease-free and overall survival following administration of FOLFOX-A for patients with resected pancreatic cancer.

DETAILED DESCRIPTION:
See summary above

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of primary pancreas invasive adenocarcinoma or adenosquamous cancer, managed with a potentially curative resection (i.e., removal of all gross tumor). Patients with invasive adenocarcinoma that also contains a component of intraductal papillary mucinous neoplasm (IPMN) are eligible.
* Interval between definitive tumor-related surgery and registration between 21-70 days.
* Patients will be staged according to the 6th edition AJCC staging system with pathologic stage T1-3, N0-1, M-0 being eligible.
* Post resection serum CA19-9 ≤ 180 units/mL within 21 days of registration on study.
* Preexisting neuropathy < grade 1 (per CTCAE).
* ECOG performance status 0 or 1.
* Age ≥ 18
* Not pregnant and not nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to beginning of treatment. Post-menopausal women (surgical menopause of lack of menses >12 months) do not need to have a pregnancy test, please document status.
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment.
* Required Initial Laboratory Values:

  * Neutrophils ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Creatinine ≤ 1.5 mg/dL -or- creatinine clearance ≥ 60 mL/min
  * Total bilirubin ≤ 1.5 x ULN
  * AST (SGOT) & ALT (SGPT) ≤ 2.5 x ULN
  * Alkaline phosphatases < 2.5x ULN
* Abdominal CT scan with contrast and chest CT/x-ray (CT of chest preferred) within 6 weeks of registration on study. Patients can have PET/MRI of the chest/abdomen instead.

Exclusion Criteria:

* Patients with serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive FOLFOX-A
* Prior hypersensitivity to Oxaliplatin or Abraxane that in the investigators opinion would put the patient at risk if re-exposed
* Patients with islet cell (neuroendocrine) tumors, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct, and ampullary carcinomas.
* Prior systemic chemotherapy for pancreas cancer; note that prior chemotherapy for a different cancer is allowable. Patients must not have received chemotherapy for a year prior to registering on study
* No prior invasive malignancy within the prior two years. However, patients with an early stage malignancy that is not expected to require treatment in the next 2 years (such as early stage, resected breast cancer or asymptomatic prostate cancer) are eligible. This must be documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — BrUOG
Locations (2):
- United States (2):
  - Roxanne Wood, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FOLFOXA
Started | 25
Completed | 24
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOXA
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 60 [43 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Adjuvant FOLFOX-A
Description: Determination of the feasibility of administration of adjuvant FOLFOX-A in patients who have undergone resection of pancreatic cancer.Successful administration of FOLFOX-A will be defined as the ability to receive ≥8 cycles of FOLFOX-A.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOXA
Number analyzed (Participants) | 24
Participants | 18

2. Secondary Outcome: Disease-free Survival
Description: To evaluate the disease-free survival for patients with resected pancreatic cancer treated with adjuvant FOLFOX-A.
Time Frame: Through study completion, an average of 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOXA
Number analyzed (Participants) | 24
Participants
  6 months after completion of drug | 23
  12 months after completion of drug | 15
  24 months after completion of drug | 12
  36 months after completion of drug | 8

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | FOLFOXA
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOXA (N=25)
Pain (General disorders) | 1 (1) — Left Hip
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXA (N=25)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 15
Infusion related reaction (Injury, poisoning and procedural complications) | 4 — Reaction to Oxaliplatin
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 14
Alanine aminotransferase increased (Investigations) | 9
Amnesia (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 13
Anorexia (Metabolism and nutrition disorders) | 6
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 9
Bloating (Gastrointestinal disorders) | 2
Blurred vision (Eye disorders) | 1
Chills (General disorders) | 3
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 10
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Edema (General disorders) | 4
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 18
Flatulence (Gastrointestinal disorders) | 4
Gait disturbance (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 14
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infections and infestations (Infections and infestations) | 8
Insomnia (Psychiatric disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 14
Lymphocyte count decreased (Investigations) | 8
Mucositis (Gastrointestinal disorders) | 9
Musculoskeletal and Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 4
Nail discoloration (Skin and subcutaneous tissue disorders) | 3
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Pain (General disorders) | 9
Platelet count decreased (Investigations) | 10
Presyncope (Nervous system disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 21
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Urinary urgency (Renal and urinary disorders) | 2
Vomitting (Gastrointestinal disorders) | 8
White blood cell decreased (Investigations) | 10
Weight loss (Investigations) | 14
Wound complication (Injury, poisoning and procedural complications) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Flu like symptoms (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02022033/Prot_SAP_ICF_000.pdf